CLINICAL TRIAL: NCT04213573
Title: Parental Perception of Silver Diamine Fluoride Staining and Its Efficacy on Caries Arrestment in Comparison to Sodium Fluoride With Casein Phosphopeptide-amorphous Calcium Phosphate
Brief Title: Efficacy of Silver Diamine Fluoride and Its Parental Perception
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: because of corona virus epidemic
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Khammas, principle investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMKhammas
Record Dates: First submitted 2019-12-18; First posted 2019-12-30 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: topical application of silver diamine fluoride (Experimental): 38% silver diamine fluoride liquid
  Interventions: Drug: silver diamine fluoride
- Group 2: topical application of MI varnish. (Active Comparator): MI Varnish:5% sodium fluoride varnish which also contains RECALDENT™* (CPP-ACP): Casein Phosphopeptide-Amorphous Calcium Phosphate
  Interventions: Drug: MI Varnish

INTERVENTIONS:
Drug: silver diamine fluoride — 38% silver diamine fluoride liquid will be applied with a brush
  Other Names: SDF
  Arms: Group 1: topical application of silver diamine fluoride
Drug: MI Varnish — topical fluoride varnish with calcium and phosphate
  Arms: Group 2: topical application of MI varnish.

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of two topical fluoride application protocols, namely 38% silver diamine fluoride and sodium fluoride with added casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) in arresting dental caries in children.

DETAILED DESCRIPTION:
The present randomized clinical study is aiming to evaluate the effectiveness of silver diamine fluoride (SDF) in arresting dentin caries lesions when compared to MI Varnish a 5% sodium fluoride varnish which also contains RECALDENT™* (CPP-ACP): Casein Phosphopeptide-Amorphous Calcium Phosphate. For this, healthy children aged 4-8 years with at least one active dentin carious lesion will be allocated randomly to one of two treatment groups: Group (1) SDF and Group (2) MI Varnish. Each participant will be assigned to one treatment group to avoid the possible synergistic effect of the different agents.

Parents/ guardians of each child will be fully informed regarding the study design, objectives and probable advantages and side effects especially the black discoloration of SDF before their involvement by written consent. The International Caries Detection and Assessment System (ICDAS II) will be used to determine caries diagnosis and activity.visual and tactile examination will be done with a WHO probe to assess the primary outcome. the secondary outcome will be conducted by a questionnaire given to the parents.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy children without any systemic disease ASA 1 physical status.
2. Children with at least one carious dentin lesion in their primary teeth, code 5 (ICDAS II)

Exclusion Criteria:

1. Children who suffer from major systemic diseases and require long term medications.
2. Children refuse the study intervention.
3. Children with silver or milk product sensitivity.
4. Presence of any gingival or perioral ulceration or stomatitis.
5. Tooth with abscess, fistula or severe pain.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
caries arrestment | 2 weeks
  The measure will be done using international caries detection and assessment system II (ICDAS II) criteria for diagnosing active and arrested caries by WHO probe

SECONDARY OUTCOMES:
Parent perception | 0 - 2 weeks
  parental perception for silver diamine fluoride staining will be conducted by questionnaire given to the parents

CONTACTS AND LOCATIONS:
Locations (1):
- al-Ameriya dental specialized center, Baghdad, Al-karkh, Iraq

IPD SHARING:
Plan to Share IPD: Undecided